CLINICAL TRIAL: NCT04833452
Title: Comparative Study Between Wide and Narrow Fenstrum Endoscopic DCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Essam Ahmed EL-mezien, Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endoscopic DCR
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Epiphora; Dacryocystitis; Dacryocystocele
Keywords: Endoscopic DCR
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Dacryocystitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide fenstrum Endoscopic DCR (Active Comparator)
  Interventions: Procedure: Endoscopic dacryocystorhinostomy
- Narrow Fenstrum Endoscopic DCR (Active Comparator)
  Interventions: Procedure: Endoscopic dacryocystorhinostomy

INTERVENTIONS:
Procedure: Endoscopic dacryocystorhinostomy — Endoscopic DCR

SUMMARY:
The aim of the study is to compare the efficacy and effectiveness of Endoscopic Endonasal DCR with narrow fenstrum approach and Endoscopic Endonasal DCR with wide fenstrum approach .

DETAILED DESCRIPTION:
The lacrimal sac and the nasolacrimal duct are contiguous structures . The part of the sac superior to the medial canthal tendon (MCT) is called the fundus, with its vertical length being 3-5 mm . The body of the sac, inferior to the MCT, is about 10 mm in length. The lacrimal sac fossa comprises of the anterior frontal process of the maxillary bone and the posterior lacrimal bone .

Lacrimal clearance relies on several factors, such as gravity, capillary attraction forces, evaporation, absorption by the conjunctival surface and the lacrimal "pump" which relies on the action of the orbicularis oculi muscle, particularly its deeper part (Horner's muscle). During the eye closing, the Horner's muscle contracts and the temporal four-fifths part of the canaliculus is pressed and closed, the nasal one-fifth part is pulled posteriorly and opens with shortening of the canalicular length. Therefore, the lacrimal fluid is effectively transported from temporal to nasal sides, finally reaching the lacrimal sac cavity. During the eye opening, as the Horner's muscle relaxes, the temporal four-fifths part of the canaliculus is expanded and the nasal one-fifth part is pressed and closed. The upper part of the lacrimal sac is directly affected by the Horner's muscle movement. During eye closing the sac expands temporally, during the eye opening the sac shrinks with an additional help of its elasticity.

The clinical evaluation of the lacrimal drainage system was originally outlined by Lester Jones. Evaluation was in the form of a dye disappearance test followed by a Jones I and Jones II test. The dye disappearance test (DDT) is useful for assessing the presence or absence of adequate lacrimal outflow, especially in unilateral cases. Using a drop of sterile 2% fluorescein solution or a moistened fluorescein strip, the examiner instills fluorescein into the conjunctival fornices of each eye and then observes the tear film.

Endoscopic DCR is a widely accepted treatment option for epiphora and dacryocystitis. endoscopic DCR has been widely performed as it has several advantages over external DCR including the absence of face scarring and better visualization via endoscopy. The purpose of DCR is to create a bypass, a rhinostoma, between the lacrimal sac and the nasal cavity.

Obstruction site in the lacrimal system is one of the characteristics contributing to a poor prognosis. False localization of the lacrimal sac and inadequate removal of the medial wall of the sac are the most common causes of failure . A systematic review showed that there was a trend towards improved outcomes and reduced granulation without increased complication rates in groups where nasal mucosal and lacrimal flaps were preserved. A study reviewing 100 failed DCR patients showed that inadequate osteotomy, incomplete sac marsupialization, and cicatricial closure of the ostium were the most common causes of failure.

To avoid or prevent obstruction of the neo-ostium, many modified techniques have been attempted. These include complete separation of the sac from the nasolacrimal duct to divert lacrimal flow to the neo-ostium, use of steroids or mitomycin-C , silicon tubing and use of mucosal flaps after wide resection of bone surrounding the sac .

Initially, endoscopic DCR relied on the creation of a relatively small fenstrum into the lacrimal sac, with the surgeon opening only the lower half of the sac. Many authors claim that the axilla of the middle turbinate is a landmark for the roof of the lacrimal sac. However, Wormald and co-authors, in a study with 47 CT-DCG patients, showed that the major part of the lacrimal sac (10 mm) is situated above the axilla of the middle turbinate, extending 1-2 mm below this landmark.

Obtaining a large marsupialized lacrimal sac with wide removal of the covering bone, medial wall of the sac and use of mucosal flaps yields a good surgical result that is comparable to the results of conventional endoscopic DCR techniques with two advantages first, primary surgical failures are amenable to technically simple and highly successful surgical revisions, second, there is a possibility for obtaining wide fenstrum without silicone tube stenting.

Success after lacrimal surgery is ill defined, and this has led to confusion in the interpretation of results for various surgical methods. The most practical measure of success is the control of symptoms, although this can be at odds with anatomic outcome.

Subjective success in turn can be assessed from the patients' symptoms. Complete relief or significant improvement of complaints can be considered a subjective success.

Anatomical patency can readily be judged in objective tests: functional endoscopic dye test or inspection of the ostium, irrigation or fluorescein retention test. Functional NLDO was first described by Demorest and Miller in 1955 to encompass lacrimal drainage dysfunction in the presence of anatomical patency. In those cases, there is a need to exclude other conditions causing epiphora, such as hyper-secretion, lacrimal pump failure, discontinuous drainage apparatus and partial lacrimal duct obstruction. The anatomical success rate i.e. the patency is reported to be higher than the functional success, which highlights the importance of measuring the physiological success and there relief of the patient's symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presented with epiphora due to nasolacrimal duct obstruction with patent canaliculi.
2. failed conservative treatment in the form of systemic antibiotics, steroid/antibiotic eye drops, decongestant nasal drops and local nasal steroid spray.
3. fit for surgery under general anesthesia.

Exclusion Criteria:

1- Epiphora due to pre-saccal obstruction of lacrimal drainage system.

2. Eye disease causing increased lacrimation and eyelid malposition

3. Lacrimal fistula.

4. Tumors of the lacrimal passage, nose or paranasal sinus.

5. Patients with abnormal bleeding or coagulation time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-08-18 (Estimated); Study Completion 2021-10-18 (Estimated)

PRIMARY OUTCOMES:
Endoscopic assessment | 1 year postoperative
  Measurement dimensions of the DCR ostium by measuring length and width in mile meters by using nasal endoscope
Objective assessment | 1 year postoperative
  Objective assessment by flourscine disappearance test

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed ragab, Cairo, Egypt

REFERENCES:
- [Background] Bertaux PJ, Gan G, Hirtz G, Mouret P, El-Hachem F, Lhuillier L, Perone JM. Evaluation of ostium size following endoscopic dacryocystorhinostomy as a predictive factor of outcome: A prospective study. J Fr Ophtalmol. 2021 Mar;44(3):397-403. doi: 10.1016/j.jfo.2020.05.024. Epub 2020 Dec 30. PMID 33388192
- [Background] Ali MJ, Psaltis AJ, Wormald PJ. Dacryocystorhinostomy ostium: parameters to evaluate and DCR ostium scoring. Clin Ophthalmol. 2014 Dec 9;8:2491-9. doi: 10.2147/OPTH.S73998. eCollection 2014. PMID 25525327
- [Background] Mann BS, Wormald PJ. Endoscopic assessment of the dacryocystorhinostomy ostium after endoscopic surgery. Laryngoscope. 2006 Jul;116(7):1172-4. doi: 10.1097/01.mlg.0000218099.33523.19. PMID 16826055